CLINICAL TRIAL: NCT00223275
Title: Naltrexone for Bipolar Disorder and Alcohol Dependence
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: E. Sherwood Brown, UT Southwestern Medical Center at Dallas
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PA-03-107
Record Dates: First submitted 2005-09-15; First posted 2005-09-22 (Estimated); Last update posted 2011-05-24 (Estimated); Status verified 2011-05

CONDITIONS: Bipolar Disorder; Alcohol Dependence
Keywords: Bipolar Disorder; Alcohol Dependence; Dual Diagnosis; Naltrexone
MeSH Terms: conditions — Bipolar Disorder; Alcoholism | interventions — Naltrexone

INTERVENTIONS:
Drug: Naltrexone

SUMMARY:
The abuse of alcohol is especially common in people with bipolar disorder. However, very little is known about how to treat people with both bipolar disorder and alcohol abuse/dependence. The purpose of this research is to determine whether naltrexone add-on therapy is associated with a greater reduction in alcohol use and alcohol craving than with placebo (an inactive substance) therapy.

DETAILED DESCRIPTION:
A 12-week, randomized, double-blind, parallel-group, placebo-controlled trial of naltrexone will be conducted in 50 English- or Spanish-speaking outpatients with bipolar I disorder or II disorder and current alcohol dependence. At the baseline appointment, informed consent will be obtained, and assessment procedures, including a review of inclusion and exclusion criteria, will be performed. The SCID (Structured Clinical Interview for DMS-IV Axis I Disorders will be performed to establish the diagnoses of bipolar I or II disorder and alcohol dependence. A psychiatrist will confirm the SCID diagnoses obtained by the RA. Eligible participants will then be given the Hamilton Rating Scale for Depression 17-item version (HRSD17), Inventory of Depressive Symptomatology-Self-Report 30-item version (IDS-SR30), Young Mania Rating Scale (YMRS), Penn Alcohol Craving Scale (PACS), Addiction Severity Index (ASI), Psychobiology of Recovery in Depression III Somatic Symptom Scale (PRD-III), and a urine drug screen. Recent alcohol use (and if present other substance use) will be assessed using the Timeline Followback (TLFB) method, with a drink defined as 13.6g of absolute alcohol (approximately 12 oz (341 mL) of beer, 5 oz of wine, 3 oz of fortified wine, or 1.5 oz of 80 proof liquor). Length of problem alcohol use will be assessed by asking, "When did alcohol first start causing you problems?" Blood will be drawn for routine laboratory analyses including a complete blood count (CBC) and SMA-20 (includes a liver panel with GGT, AST, ALT, Billirubin) at baseline (week 0) and completion (week 12). Blood will also be drawn at weeks 4 and 8 for repeat testing of GGT levels. A physical examination will be performed at baseline. Women of childbearing potential will receive a urine pregnancy test and will be counseled about effective contraceptive methods. A psychiatrist will assess the participants at baseline and weekly follow-up visits, and will participate in the informed consent process. Study medication will be given at a second appointment after results of the liver function tests have been received (generally 1-2 days after the first appointment). At each weekly assessment the HRSD17, IDS-R30, YMRS, an assessment of alcohol use in the past week, and a urine drug screen will again be obtained. Urine drug screen will be obtained only from the newly enrolled subjects. We will not obtain urine drug screens from subjects who are already active in the study. In addition, all participants will receive a total of 16 one-hour/week sessions of manual-driven CBT specifically designed for persons with bipolar disorder and substance abuse, provided by a bilingual psychologist with experience in CBT. Patients will discontinue study medication at week 12, but continue their CBT therapy until week 16. Pill counts will be conducted at each weekly assessment visit. In addition, during weekly assessments, participants will be asked about adherence with other psychotropic medications using a modified version of an assessment developed by Weiss et al., and the estimated percent of prescribed medication actually taken will be recorded.

ELIGIBILITY:
INCLUSION CRITERIA:

* English or Spanish-speaking
* Age 18-70
* Diagnosis of bipolar I or II.
* Current mood state of depressed or mixed.
* Alcohol use of at least 5 drinks in the past 7 days.
* Current diagnosis of alcohol dependence.

EXCLUSION CRITERIA:

* Bipolar disorders other than bipolar I or II disorders (e.g., bipolar NOS, or cyclothymic disorders, schizophrenia, schizoaffective disorder, or unipolar).
* Lifetime opiate abuse or dependence or any current use (including prescription drugs).
* Diagnosis of current dependence on substances other than alcohol (participants with only abuse of other substances are included. Dependence on caffeine and/or nicotine is allowed.)
* Severe or life-threatening medical illness (e.g., hepatic cirrhosis, congestive heart failure, terminal cancer) or labs consistent with serious medical illness (e.g., severe edema, atrial fibrillation, dangerously abnormal electrolytes).
* Pregnant or nursing female
* High risk for suicide defined as ≥2 suicide attempts in the past 12 months that required medical attention, or current suicidal ideation with plan and intent.
* Prior therapy with naltrexone and/or allergic reaction to naltrexone.
* Current therapy with acamprosate or disulfiram.
* Member of a vulnerable population (Dementia, cognitively impaired, mental retardation, prisoner)
* Baseline YMRS or HRSD17 scores ≥ 30.
* AST, ALT, or bilirubin > 3 times upper limit of normal.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2005-05; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edson S Brown, MD, PhD, Principal Investigator — UT Southwestern Medical Center Dallas
Locations (1):
- UTSouthwestern Medical Center, Dallas, Texas, United States